CLINICAL TRIAL: NCT06407921
Title: Comparative Effects of Whole Body Vibration and BOSU Ball on Balance and Functional Mobility in Children With Spastic Cerebral Palsy
Brief Title: Whole Body Vibration and BOSU Ball in Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/07100
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Spastic Cerebral Palsy
Keywords: cerebral palsy; WBVT; bosu ball; functional mobility; balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: It will be randomized control trial in which non probability convenient sampling will be used. Two groups of 6-12 age will be formed in which participants will be randomly divided. group A will only receive Whole Body Vibration therapy and group B will only receive BOSU ball.
Who Masked: Participant
Masking Description: Participant's will get separate treatment protocols and possible efforts will be put to msk the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Body Vibration Therapy (Experimental): This group will receive Whole Body Vibration Therapy
  Interventions: Device: Whole Body Vibration
- BOSU ball therapy (Experimental): This group will receive BOSU ball therapy
  Interventions: Device: BOSU ball

INTERVENTIONS:
Device: Whole Body Vibration — On vibration plate pate child will do kneeling, and one leg standing, standing horizontally or vertically. Along routine physical therapy such as stretching activities to keep up muscle elasticity particularly Achilles tendon, hamstring muscles, hip flexors and adductors, shoulder internal rotators, elbow and wrist flexors, pronators, and ulnar deviators, each stretch will be given for 30 seconds with 3 repetitions.Strength training to hip flexor, knee extensor, and ankle dorsiflexors for 15 minutes 3 times a week for 8 weeks. Session will be of 30 minutes
  Arms: Whole Body Vibration Therapy
Device: BOSU ball — Exercises such as (1) standing on a BOSU ball while throwing and catching a ball (2) 1-legged standing (affected leg) on the BOSU ball while throwing and catching a ball with therapist support; and (3) small jumps on the BOSU ball. Three sets of 6 repetitions for each exercise will be perform every 2 weeks up to a maximum of 10 repetitions if the participants were still able to perform the training easily. Total dose of balance training in 1 session will be 15 minutes
  Arms: BOSU ball therapy

SUMMARY:
Cerebral palsy is a non-progressive neurodevelopmental disorder, also known as littles disease. The most common cause of physical and mental disabilities in the pediatric population. Cerebral means brain and palsy means weakness or problems in muscles. Spastic cerebral palsy is the common type of cerebral palsy characterized by spasticity or high muscle tone, results in stiffness etc.

This will be a randomized clinical trial, data will be collected from Sehat medical complex Lahore. Study will be conducted on 30 patients. Inclusion criteria of this study is spastic diplegic CP children with age between 6 to 12 years, with GMFCS level 1 and 2 and those both male nd female, able to understand command will be included. Those diplegic spastic CP who have orthopedic intervention/surgery, botulinum toxin injection within past six months, or medical problems such as pneumonia that prevented children from participating in exercises will be excluded.

DETAILED DESCRIPTION:
Group A: whole body vibration therapy group This group will be provided with whole body vibration therapy in spastic cerebral palsy children. Exercise will be conducted 3 times a week for 8 weeks. Pre and post session functional mobility and balance will be measured by pediatric balance scale and time up and go test. Along routine physical therapy such as stretching exercise of achilles tendon, hamstring muscles, hip flexors and adductors, shoulder internal rotators, and wrist flexors, pronators, and ulnar deviator etc.

Group B: BOSU ball training group This group will be provided with both sides up ball BOSU training in spastic cerebral palsy children. Exercise will be conducted 3 times a week for 8 weeks. Pre and post session functional mobility and balance will be measured by pediatric balance scale and time up and go test. Along routine physical therapy such as stretching exercise of achilles tendon, hamstring muscles, hip flexors and adductors, shoulder internal rotators, and wrist flexors, pronators, and ulnar deviator etc.

ELIGIBILITY:
Inclusion Criteria:

* Spastic diplegic CP with GMFCS level I-II
* Age 6-12 years
* Both male and female.
* Able to understand command

Exclusion Criteria:

* Orthopedic surgery within 6 months
* Botulinum injection
* Parents refuse to participate
* Other diseases as Pneumonia

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale | 8 weeks
  The (PBS) pediatric balance scale, a modification of the Berg Balance Scale, was developed as a balance measure for school-age children with mild-to-moderate motor impairments. It gives good test-retest and interrater reliability when used, ranged from 0.87 to 1.0.
Timed Up & Go test | 8 weeks
  TUG is used to determine functional mobility.Functional mobility of children will be evaluated through timed get up and go (TUG) test and its results will be recorded. In this test, the duration of standing up from the chair, walking up to 3 m, returning, and sitting on the chair will be measured. It is a very valid and reliable tool 0.97 and 0.99.
Functional Mobility Scale | 8 weeks
  FMS (functional mobility scale) is used to measure functional mobility and its results will be recorded. It has perfect test-retest reliability (κw=0.98-1.00)

CONTACTS AND LOCATIONS:
Overall Officials: Hafsa Imtiaz, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah JP, Thaker N, Heimur J, Aredo JV, Sikdar S, Gerber L. Myofascial Trigger Points Then and Now: A Historical and Scientific Perspective. PM R. 2015 Jul;7(7):746-761. doi: 10.1016/j.pmrj.2015.01.024. Epub 2015 Feb 24. PMID 25724849